CLINICAL TRIAL: NCT03251625
Title: Supplementation With a Multi-strain Probiotic Formulation (Bio-Kult®) in the Management of Diarrhea-predominant Irritable Bowel Syndrome - a Randomized, Double-blind, Placebo-controlled Clinical Trial
Brief Title: Multi-strain Probiotic in the Management of IBS-D
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh (Other)
Responsible Party: Principal Investigator, S M khosruzzaman, Principal Investigator, Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: No. BSMMU/2015/1011
Record Dates: First submitted 2017-08-09; First posted 2017-08-16 (Actual); Last update posted 2018-02-05 (Actual); Status verified 2018-02

CONDITIONS: Irritable Bowel Syndrome
MeSH Terms: conditions — Irritable Bowel Syndrome

STUDY DESIGN:
Intervention Model Description: a randomized, double-blind, placebo-controlled clinical trial
Who Masked: Participant, Investigator
Masking Description: Participants divided into two groups by randomization software, consisting of 200 in each group.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- To assess the effect of multistrain probiotics on abdominal (Placebo Comparator): To assess the effect of multistrain probiotics on abdominal pain using a validated symptom severity score in IBS patients.
  Interventions: Drug: Probiotic Formula Capsule
- To assess the efficacy of a multistrain probiotic supplement (Placebo Comparator): To assess the efficacy of a multistrain probiotic supplement as a treatment option for IBS in a tertiary referral centre
  Interventions: Drug: Probiotic Formula Capsule

INTERVENTIONS:
Drug: Probiotic Formula Capsule

SUMMARY:
1. To assess the effect of multistrain probiotics on abdominal pain using a validated symptom severity score in IBS patients.
2. To assess the efficacy of a multi-strain probiotic supplement as a treatment option for IBS in a tertiary referral centre

DETAILED DESCRIPTION:
Background: Accumulating evidence supports the view that an imbalance of gut bacteria contributes to IBS, and that increasing the mass of beneficial species may reduce the numbers of pathogenic bacteria and help alleviate symptoms.

Methods: In this double-blind trial 360 adult patients with moderate-to-severe symptomatic diarrhea-predominant IBS (IBS-D) were randomized to treatment with the multi-strain probiotic (Bio-Kult®; 14 different bacterial strains; 8 billion colony-forming units per day) or placebo for 16 weeks. The change in severity and frequency of abdominal pain was the primary outcome measure.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed case of IBS using Rome III criteria
2. Absence of red flag sign: anemia, fever, wt loss, per rectal bleeding, nocturnal frequency, family history of inflammatory bowel disease (IBD), cancer
3. Age 18-55 years
4. No probiotics used in prior 3 months.
5. Agreed not to start any other drug unless clinically indicated.
6. No antibiotics in previous 2 months of enrolment.

Exclusion Criteria:

1. Age<18 or >55 years
2. Previous treatment with probiotics within last 3 months
3. Pregnant or lactating females
4. Concurrent severe illness (Uncontrolled diabetes mellitus, Renal Dysfunction, Liver disease, hyper and hypothyroidism)
5. Chronic organic bowel disorders e.g. inflammatory bowel diseases, tuberculosis, Diverticular disease etc
6. Any previous gastrointestinal surgery

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 400 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
The change in severity and frequency of abdominal pain during treatment with a multi-strain probiotic or placebo | 1 year.
  The change in severity and frequency of abdominal pain as measured by IBS-Symptom Severity Scores during treatment with a multi-strain probiotic or placebo, and compared with baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Ashton Harper, MRCS, Study Director — Probiotics International Ltd (Protexin)

IPD SHARING:
Plan to Share IPD: Undecided
After completion of paper.

REFERENCES:
- [Derived] Ishaque SM, Khosruzzaman SM, Ahmed DS, Sah MP. A randomized placebo-controlled clinical trial of a multi-strain probiotic formulation (Bio-Kult(R)) in the management of diarrhea-predominant irritable bowel syndrome. BMC Gastroenterol. 2018 May 25;18(1):71. doi: 10.1186/s12876-018-0788-9. PMID 29801486

DOCUMENTS (1):
  • Study Protocol (2015-08-02): https://cdn.clinicaltrials.gov/large-docs/25/NCT03251625/Prot_000.pdf